CLINICAL TRIAL: NCT04182776
Title: Fragility Fractures of the Pelvis: Observational Outcome Study
Brief Title: Fragility Fractures of the Pelvis (FFP)
Status: Recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: AOFFP
Record Dates: First submitted 2019-11-25; First posted 2019-12-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pelvic Fracture
Keywords: Pelvis; Fragility Fracture; Classification; Conservative; Operative
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelvis fracture type II to IV: All treatments will remain the standard (routine) care procedures based on individual clinician's judgment and the patient characteristics. The registry does not dictate any specific treatment.

SUMMARY:
Prospective data will be collected in approximately 420 patients, above the age of 65, suffering from an FFP type fracture equal to or higher than type II, according to Rommens and Hofmann.

Patients will be followed up according to the standard (routine) for up to 1 year after the treatment. Data collection will include underlying disease, treatment details, functional and patient reported outcomes (PRO)s, radiological outcomes, and anticipated or procedure-related adverse events (i.e. complications).

DETAILED DESCRIPTION:
More in detail this registry has the following objectives:

* To identify the difference in patient related outcome comparing the surgical and conservative treatment in patients suffering from an FFP with different levels of pelvic instability at different time points
* To compare the rate of complications, morbidity and mortality between the different treatment modalities over the whole study period

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older at time of injury
* Diagnosis, via CT scan as per standard of care, of FFP grade II or higher according to the Rommens and Hofmann classification (including fractures of the anterior pelvic ring involving the anterior lip of the acetabulum not regarded as the acetabular fractures)
* Informed consent obtained, ie:

  * Ability to understand the content of the patient information/ICF
  * Willingness and ability to participate in the registry according to the standard of care in each clinic
  * Signed and dated Ethics Committee (EC)/ Institutional Review Board (IRB) approved written informed consent OR
  * Written consent provided according to the IRB/EC defined and approved procedures for patients who are not able to provide independent written informed consent

Exclusion Criteria:

* Pelvic fractures that do not meet the criteria of a fragility fracture (ie, high-energy trauma)
* FFP type I fractures
* Concomitant fractures of the acetabulum (except anterior lip of the acetabulum, see above)
* Pathological fractures (ie, patients with malignant or metastatic diseases of the pelvis, infections)
* Concomitant osteoporotic fractures outside of pelvis
* Participation in any other medical device or medicinal product study within the previous month that could influence in opinion of the PI the results of the present registry

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (over 65) who have suffered from fragility fractures of the pelvis (FFP), equal to or higher than type II (according to Rommens and Hofmann)
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Demographics | Pre-treatment
  Year of birth, Gender, Ethnicity, Height (cm) and Weight (kg) will be combined to report BMI in kg/m^2
Comorbidities | Pre-treatment
  Concomitant diseases will be assessed using the Charlson Comorbidity Index (CCI). This score assesses the comorbidity level by considering both the number and severity of pre-defined comorbid conditions. It provides a weighted score of a patient's comorbidities which can be used to predict mortality rates. It is a 17-items questionnaire with score range from 0 to 37 points. It estimates the 10-year (or shorter) patient survival.
Cognitive status | Pre-treatment
  The MiniCog is a 3-minute instrument assessing cognitive impairment. It consists of two components, a 3-item recall test for memory and a simply scored clock drawing test. A total score ranges from 0 to 5. A score of zero, one or two out of five points in total, indicates a concern in cognitive functioning.
Patient-reported outcomes: PROMIS Pain Interference | from the pre-treatment assessment until 12 months after the treatment (surgical or not-surgical)
  PROMIS (Patient-Reported Outcome Measurement Information System) Pain Interference (8 questions) assesses the impact of pain on common activities of daily life including social, cognitive, emotional, physical, and recreational aspects. The higher score represents a higher pain level.
Patient-reported outcomes: PROMIS Physical Function | from the pre-treatment assessment until 12 months after the treatment (surgical or not-surgical)
  PROMIS Physical Function (10 questions) assesses self-reported capability of physical activities including instrumental activities of daily living. A higher score indicates a better self-reported capability.
Patient Reported Outcomes - EuroQoL (EQ-5D-3L) | from the pre-treatment assessment until 12 months after the treatment (surgical or not-surgical)
  The EQ-5D-3L has five items (mobility, self-care, usual activities, pain/discomfort anxiety/depression) with a three-point categorical response scale level (1 = no problems, 2 = some / moderate problems, 3 = extreme problems) where the patient's current health status is assessed. A unique EQ-5D-3L health state is defined by combining one level from each of the five dimensions. The EQ-5D index score ranges from 0 (death) to 1 (best imaginable quality of life), and negative values express "worse than death" state.

SECONDARY OUTCOMES:
Parker Mobility Score | from the pre-treatment assessment until 12 months after the treatment (surgical or not-surgical)
  Parker Mobility Scale assess the patient's ability to perform indoor walking, outdoor walking, and shopping before the fracture. A score ranges between 0 and 3 (0 = not at all, 1 = with help from another person, 2 = with an aid, and 3 = no difficulty and no aid) for each function, resulting in a total score ranging from 0 (no walking ability at all) to 9 (fully independent).
Modified Barthel index | from the pre-treatment assessment until 12 months after the treatment (surgical or not-surgical)
  The Barthel index is an ordinal scale and each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses 10 variables describing activities of daily living and mobility. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital.
Residential status | from the pre-treatment assessment until 12 months after the treatment (surgical or not-surgical)
  The residential status will be documented at each visit during 1-year post-treatment phase.
Mortality | from the pre-treatment assessment until 12 months after the treatment (surgical or not-surgical)
  Mortality will be assessed for 4 phases:
  * Perioperative mortality
  * Within the first 7 days after treatment (early-term)
  * Within the first 3 months after treatment (mid-term)
  * Until the last follow up (long-term mortality)
Radiological outcomes | from the pre-treatment assessment until 12 months after the treatment (surgical or not-surgical)
  Position of the fracture fragments, to rule out secondary (additional) fracture fragments and displacement, or loosening of implants (Undisplaced, Displaced, Non-union with extensive callus)
Anticipated treatment or condition-related adverse events (i.e. complications) | from the pre-treatment assessment until 12 months after the treatment (surgical or not-surgical)
  In this registry, only condition- or treatment-related events (ie complications) will be collected . Partially those events presuppose themselves: eg, re-admission for a surgical revision. In those cases, details on those different events will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Pol Maria Rommens, MD, Principal Investigator — University Medical Center Johannes Gutenberg-University
Locations (10):
- University of Missouri, Columbia, Missouri, United States
- The Ottawa Hospital - Civic Campus, Ottawa, Canada
- Germany (3):
  - University Medical Center Hamburg Eppendorf, Hamburg
  - University Hospital Leipzig, Leipzig
  - University Medical Center Johannes Gutenberg-University, Mainz
- Queen Mary Hospital, Hong Kong, Hong Kong
- Okayama medical hospital, Okayama, Japan
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Radboud University Medical Center, Nijmegen
- Cantonal Hospital Lucerne, Lucerne, Switzerland